CLINICAL TRIAL: NCT04826770
Title: Blood Donations From Healthy Probands for the Study of the Adaptive Immune Response to COVID-19 Vaccination (AICOVI)
Brief Title: Adaptive Immune Response to COVID-19 Vaccination
Acronym: AICOVI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Sponsor
Other Study IDs: BB 001/21f
Record Dates: First submitted 2021-03-22; First posted 2021-04-01 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-10

CONDITIONS: SARS-CoV-2 Vaccination
Keywords: vaccine; vaccination; SARS-CoV-2; COVID-19; immune response; immunokinetics
MeSH Terms: conditions — COVID-19 | interventions — BNT162 Vaccine; ChAdOx1 nCoV-19; 2019-nCoV Vaccine mRNA-1273

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA plasma, peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- BNT/BNT/BNT: Subjects receiving two doses of BNT162b2 (Comirnaty®, tozinameran (INN), BioNTech/Pfizer) as homologous basic immunization and one dose of BNT162b2 as booster vaccination
  Interventions: Drug: BNT162b2
- AZD/BNT/BNT: Subjects receiving one dose of AZD 1222 (Vaxzevria®, Covishield®, ChadOx1 nCoV-19, Oxford University/Astra-Zeneca) followed by one dose of BNT162b2 (Comirnaty®, tozinameran (INN), BioNTech/Pfizer) as heterologous basic immunization and one dose of BNT162b2 (Comirnaty®, tozinameran (INN), BioNTech/Pfizer) as booster vaccination
  Interventions: Drug: BNT162b2; Drug: AZD 1222
- AZD/AZD/BNT: Subjects receiving two doses of AZD 1222 (Vaxzevria®, Covishield®, ChadOx1 nCoV-19, Oxford University/Astra-Zeneca) as homologous basic immunization and one dose of BNT162b2 (Comirnaty®, tozinameran (INN), BioNTech/Pfizer) as booster vaccination
  Interventions: Drug: BNT162b2; Drug: AZD 1222
- AZD/MOD/BNT: Subject receiving one dose of AZD 1222 (Vaxzevria®, Covishield®, ChadOx1 nCoV-19, Oxford University/Astra-Zeneca) followed by one dose of mRNA-1273 (Spikevax®, elasomeran (INN), Moderna) as heterologous basic immunization and one dose of BNT162b2 (Comirnaty®, tozinameran (INN), BioNTech/Pfizer) as booster vaccination
  Interventions: Drug: BNT162b2; Drug: AZD 1222; Drug: mRNA-1273
- AZD/BNT/MOD: Subject receiving one dose of AZD 1222 (Vaxzevria®, Covishield®, ChadOx1 nCoV-19, Oxford University/Astra-Zeneca) followed by one dose of BNT162b2 (Comirnaty®, tozinameran (INN), BioNTech/Pfizer) as heterologous basic immunization and one dose of mRNA-1273 (Spikevax®, elasomeran (INN), Moderna) as booster vaccination
  Interventions: Drug: BNT162b2; Drug: AZD 1222; Drug: mRNA-1273
- Control/validation group: Control samples for the validation of the used methods from the pre-SARS-CoV-2 era were transferred from the study "Blood Donations from Healthy Blood Donors to Investigate Circannual Variations in Tryptophan Metabolism and Adaptive Immune Response to Bacterial Infectious Agents" (in short TRP study). Subjects had not received any SARS-CoV-2 vaccination at that time. Remaining plasma samples were transferred to the AICOVI study.

INTERVENTIONS:
Drug: BNT162b2 — vaccination against COVID-19
  Other Names: Comirnaty®; tozinameran
  Groups: AZD/AZD/BNT; AZD/BNT/BNT; AZD/BNT/MOD; AZD/MOD/BNT; BNT/BNT/BNT
Drug: AZD 1222 — vaccination against COVID-19
  Other Names: Vaxzevria®; Covishield®; ChadOx1 nCoV-19
  Groups: AZD/AZD/BNT; AZD/BNT/BNT; AZD/BNT/MOD; AZD/MOD/BNT
Drug: mRNA-1273 — vaccination against COVID-19
  Other Names: Spikevax®; elasomeran
  Groups: AZD/BNT/MOD; AZD/MOD/BNT

SUMMARY:
AICOVI (Adaptive Immune Response to COVID-19 Vaccination) is a prospective clinical cohort study aiming at studying the kinetics of vaccine-specific antibody production after COVID-19 vaccination in health care workers.

DETAILED DESCRIPTION:
AICOVI (Adaptive Immune Response to COVID-19 Vaccination) is a prospective clinical cohort study aiming at elucidating the kinetics of vaccine-specific antibody production after COVID-19 vaccination in health care workers at the Greifswald University hospital.

Participants were recruited before their intended vaccination. Participants received the basic immunization with either two i. m. doses of BNT162b2 (Comirnaty®, tozinameran (INN), BioNTech/Pfizer) with a time interval of 21 days or two i. m. dose of AZD 1222 (Vaxzevria®, Covishield®, ChadOx1 nCoV-19, Oxford University/Astra-Zeneca) with a time interval of 12 weeks (homologous vaccination), or one i. m. dose of AZD 1222 as the first vaccination and one i. m. dose of BNT162b2 or mRNA-1273 (Spikevax®, elasomeran (INN), Moderna) as the second vaccination with a time interval of at least 4 weeks (heterologous vaccination). Approximately 6 months later, participants received a booster vaccination with BNT162b2.

Within the study, volunteers donate peripheral blood by venipuncture on each day of vaccination as well as 7 and 14 days after each vaccination. EDTA plasma and peripheral mononuclear cells (PBMCs) are prepared and stored at -20 °C.

Volunteers are also asked to complete a standardized questionnaire on each day of blood sampling. Questionnaires collect data about physical characteristics, COVID-19 vaccination, previous SARS-CoV-2 infection as well as current infections, medication, immune relevant diseases and side effects of the vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Planned participation in COVID-19 vaccination
* Completion of the 18th year of life
* verbal and written consent given

Exclusion Criteria:

* current infectious diseases
* underweight (BMI<18,5)
* blood coagulation disorders, anemia or similar diseases
* known congenital or acquired immunodeficiencies

Inclusion criteria for control/validation group of TRP participants:

* informed written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Employees at the University Medicine Greifswald, Germany, who plan to be vaccinated against COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-01-06 (Actual); Primary Completion 2021-12-13 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
mean current anti-SARS-CoV-2 antibody production and cumulative antibody titer on the day of the 1st vaccination | 1 day
  Serum antibody titers represent a cumulative measure of any preceded or recent immune responses. The current antibody production can be quantified using MENSA (medium enriched for newly synthesized antibodies), an approach that measures antibodies released from recently stimulated circulating antibody-secreting plasmablasts. For this purpose PBMCs are collected from the subject's whole blood sample, washed to remove serum antibodies, and then cultured for 7 days. Antibodies released ex vivo from the antibody-secreting plasmablasts can now be detected in the culture supernatant. These newly synthesized antibodies are a measure of the instantaneous antibody response.
  Sampling is conducted on the day of the 1st vaccination.
mean current anti-SARS-CoV-2 antibody production 7 days after the 1st vaccination | 7 days after the 1st vaccination
  Serum antibody titers represent a cumulative measure of any preceded or recent immune responses. The current antibody production can be quantified using MENSA (medium enriched for newly synthesized antibodies), an approach that measures antibodies released from recently stimulated circulating antibody-secreting plasmablasts. For this purpose, PBMCs are collected from the subject's whole blood sample, washed to remove serum antibodies, and then cultured for 7 days. Antibodies released ex vivo from the antibody-secreting plasmablasts can now be detected in the culture supernatant. These newly synthesized antibodies are a measure of the instantaneous antibody response.
  Sampling is conducted 7 days after the 1st vaccination.
mean current anti-SARS-CoV-2 antibody production 14 days after the 1st vaccination | 14 days after the 1st vaccination
  Serum antibody titers represent a cumulative measure of any preceded or recent immune responses. The current antibody production can be quantified using MENSA (medium enriched for newly synthesized antibodies), an approach that measures antibodies released from recently stimulated circulating antibody-secreting plasmablasts. For this purpose, PBMCs are collected from the subject's whole blood sample, washed to remove serum antibodies, and then cultured for 7 days. Antibodies released ex vivo from the antibody-secreting plasmablasts can now be detected in the culture supernatant. These newly synthesized antibodies are a measure of the instantaneous antibody response.
  Sampling is conducted 14 days after the 1st vaccination.
mean current anti-SARS-CoV-2 antibody production on the day of the 2nd vaccination | day of the 2nd vaccination
  Serum antibody titers represent a cumulative measure of any preceded or recent immune responses. The current antibody production can be quantified using MENSA (medium enriched for newly synthesized antibodies), an approach that measures antibodies released from recently stimulated circulating antibody-secreting plasmablasts. For this purpose, PBMCs are collected from the subject's whole blood sample, washed to remove serum antibodies, and then cultured for 7 days. Antibodies released ex vivo from the antibody-secreting plasmablasts can now be detected in the culture supernatant. These newly synthesized antibodies are a measure of the instantaneous antibody response.
  Sampling is conducted on the day of the 2nd vaccination.
mean current anti-SARS-CoV-2 antibody production 7 days after the 2nd vaccination | 7 days after the 2nd vaccination
  Serum antibody titers represent a cumulative measure of any preceded or recent immune responses. The current antibody production can be quantified using MENSA (medium enriched for newly synthesized antibodies), an approach that measures antibodies released from recently stimulated circulating antibody-secreting plasmablasts. For this purpose, PBMCs are collected from the subject's whole blood sample, washed to remove serum antibodies, and then cultured for 7 days. Antibodies released ex vivo from the antibody-secreting plasmablasts can now be detected in the culture supernatant. These newly synthesized antibodies are a measure of the instantaneous antibody response.
  Sampling is conducted 7 days after the 2nd vaccination.
mean current anti-SARS-CoV-2 antibody production 14 days after the 2nd vaccination | 14 days after the 2nd vaccination
  Serum antibody titers represent a cumulative measure of any preceded or recent immune responses. The current antibody production can be quantified using MENSA (medium enriched for newly synthesized antibodies), an approach that measures antibodies released from recently stimulated circulating antibody-secreting plasmablasts. For this purpose, PBMCs are collected from the subject's whole blood sample, washed to remove serum antibodies, and then cultured for 7 days. Antibodies released ex vivo from the antibody-secreting plasmablasts can now be detected in the culture supernatant. These newly synthesized antibodies are a measure of the instantaneous antibody response.
  Sampling is conducted 14 days after the 2nd vaccination.
mean current anti-SARS-CoV-2 antibody production and cumulative antibody titer on the day of the booster vaccination | 1 day
  Serum antibody titers represent a cumulative measure of any preceded or recent immune responses. The current antibody production can be quantified using MENSA (medium enriched for newly synthesized antibodies), an approach that measures antibodies released from recently stimulated circulating antibody-secreting plasmablasts.
  For this purpose PBMCs are collected from the subject's whole blood sample, washed to remove serum antibodies, and then cultured for 7 days. Antibodies released ex vivo from the antibody-secreting plasmablasts can now be detected in the culture supernatant. These newly synthesized antibodies are a measure of the instantaneous antibody response.
  Sampling is conducted on the day of the booster vaccination.
mean current anti-SARS-CoV-2 antibody production 7 days after the booster vaccination | 7 days after the booster vaccination
  Serum antibody titers represent a cumulative measure of any preceded or recent immune responses. The current antibody production can be quantified using MENSA (medium enriched for newly synthesized antibodies), an approach that measures antibodies released from recently stimulated circulating antibody-secreting plasmablasts. For this purpose, PBMCs are collected from the subject's whole blood sample, washed to remove serum antibodies, and then cultured for 7 days. Antibodies released ex vivo from the antibody-secreting plasmablasts can now be detected in the culture supernatant. These newly synthesized antibodies are a measure of the instantaneous antibody response.
  Sampling is conducted 7 days after the booster vaccination.
mean current anti-SARS-CoV-2 antibody production 14 days after the booster vaccination | 14 days after the booster vaccination
  Serum antibody titers represent a cumulative measure of any preceded or recent immune responses. The current antibody production can be quantified using MENSA (medium enriched for newly synthesized antibodies), an approach that measures antibodies released from recently stimulated circulating antibody-secreting plasmablasts. For this purpose, PBMCs are collected from the subject's whole blood sample, washed to remove serum antibodies, and then cultured for 7 days. Antibodies released ex vivo from the antibody-secreting plasmablasts can now be detected in the culture supernatant. These newly synthesized antibodies are a measure of the instantaneous antibody response.
  Sampling is conducted 14 days after the booster vaccination.

SECONDARY OUTCOMES:
plasma antibody levels against SARS-CoV-2 | On each day of vaccination as well as 7 and 14 days after each vaccination
  Anti-SARS-CoV-2 antibodies are quantified using ELISA and/or xMAP(R) technology.
immune cell phenotyping (B cells, T cells) | On each day of vaccination as well as 7 and 14 days after each vaccination
  flow cytometry-based analyses
Characterization of antibody proteomics profile changes after vaccination | On each day of vaccination as well as 7 and 14 days after each vaccination
  The antibody profile in plasma is assessed using mass spectrometry.
Characterization of the cytokine profile elicited after vaccination | On each day of vaccination as well as 7 and 14 days after each vaccination
  The cytokine profile elicited after vaccination is assessed using a multiplex immunoassay.
Measurement of neutralizating antibodies after vaccination | On each day of vaccination as well as 7 and 14 days after each vaccination
  Neutralizing antibodies are measured by neutralization tests.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara M. Bröker, Prof. Dr., Study Chair — University Medicine Greifswald, Dept. of Immunology
Locations (1):
- University Medicine Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: Undecided